CLINICAL TRIAL: NCT02944812
Title: Chidamide for Refractory/Relapsed Peripheral T Cell Lymphoma, a Single-Center, Nonrandomized Phase II Clinical Trial
Brief Title: Chidamide for Refractory/Relapsed Peripheral T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wenyu Li, Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WYli-002
Record Dates: First submitted 2016-10-21; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide (Experimental): Chidamide is given to the patients, the dosage is 30mg,biw,po.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide is given to the patients as described, and drug concentration is measured in patients' serum and CSF, also, parameters concerning efficacy and safety are also obtained.
  Other Names: epidaza

SUMMARY:
This trial intends: 1.To evaluate the concentration of Chidamide in the serum and cerebral-spinal fluid of PTCL patients at certain time points after taking the medicine, to evaluate the pharmacokinetics of Chidamide in these patients and its CNS (central nervous system) distribution.

2. To evaluate the efficiency and safety of Chidamide in PTCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. PTCL patients confirmed by histopathology examination.
2. Did not accept radiotherapy, chemotherapy, targeted-therapy or hematopoietic stem cell transplantation within 4 weeks prior to inclusion;
3. Age 18-75 years old, male or female;
4. ECOG: 0-1 point;
5. Body weight: male 67±20 kilograms (47-87 kg), female 55±20 kilograms (35-75 kg);
6. Blood-routine test should satisfy (except lymphoma-related abnormalities): Hb≥90g/L，ANC≥1.5×109/L，PLT≥90×109/L；
7. Estimated survival ≥ 3 months;
8. Willing to sign the written consent before the trial.

Exclusion Criteria:

1. Women during pregnancy or lactation, or fertile women unwilling to take contraceptive measures.
2. QTc elongation with clinical significance (˃ 480ms), ventricular tachycardia, atrial fibrillation, cardiac conducting blockage, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease that requires treatment.
3. Cardiac B ultrasound show end-diastolic pericardial dark zone≥ 10mm
4. Patients who have received organ transplantation.
5. Patients received symptomatic treatment for bone marrow toxicity within 7 days prior to enrollment.
6. Patients with active hemorrhage.
7. Patients with or with history of thrombosis, embolism, cerebral hemorrhage, or cerebral infarction.
8. Patients with active infection, or with continuous fever within 14 days prior to enrollment.
9. Had major organ surgery within 6 weeks prior to enrollment.
10. Impaired liver function ( Total bilirubin ˃ 1.5 times of normal maximum, ALT/AST˃ 2.5 times of normal maximum, for patients with infiltrative liver disease ALT/AST ˃ 5 times of normal maximum), impaired renal function (serum creatinin˃ 1.5 times of normal maximum).
11. Patients with mental disorders or those do not have the ability to consent;
12. Patients with drug abuse, long term alcoholism that may impact the results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change of Chidamide concentration within the serum | 5 minutes before taking Chidamide (0h) and 1h, 2h, 4h, 8h and 12h after taking Chidamide (1h，2h，4h，8h，12h), assessed up to 1 week from date of enrollment.
Change of Chidamide concentration within the cerebral-spinal fluid (CSF) | 5 minutes before the first dosage of Chidamide (0h) and 4 hours after the second dosage (4h) of Chidamide

SECONDARY OUTCOMES:
white blood cell count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
red blood cell count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood Hb level | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood platelet count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
vital signs | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum alanine aminotransferase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum aspartate transaminase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum total bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum direct bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum indirect bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum glutamyltranspeptidase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum albumin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum ureal nitrogen level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum creatinin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood electrolytes level（K+, Na+，Cl-，Ca2+，Mg2+） | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood LDH level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
QTc from ECG | every 6 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong general hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Data of the trial would be available on the corresponding website after the trial has been finished.